CLINICAL TRIAL: NCT06602739
Title: A Randomized, Double-Masked, Placebo-Controlled Study to Assess the Efficacy and Safety of REGN5713-5715 to Reduce Signs and Symptoms of Allergic Conjunctivitis in Participants With Birch Pollen Allergy
Brief Title: A Study to Demonstrate the Effect of REGN5713-5715 on Reducing Ocular Allergy Signs and Symptoms in Adult Participants With Birch Pollen Allergy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R5713-5715-ALG-2415
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Allergic Conjunctivitis
Keywords: Birch Pollen Allergy; Ocular allergy symptoms; Ocular allergy signs
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- REGN5713-5715 (Experimental): Participants will be randomized 1:1
  Interventions: Drug: REGN5713; Drug: REGN5715
- Placebo (Placebo Comparator): Participants will be randomized 1:1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REGN5713 — Administered per protocol
  Other Names: Bremzalerbart
  Arms: REGN5713-5715
Drug: REGN5715 — Administered per protocol
  Other Names: Atisnolerbart
  Arms: REGN5713-5715
Drug: Placebo — Administered per protocol
  Arms: Placebo

SUMMARY:
This study is researching 2 experimental drugs, REGN5713 and REGN5715, which are called REGN5713-5715 when mixed together (called "study drug") to reduce eye allergy signs and symptoms due to birch tree pollen allergy.

The aim of the study is to see how safe and effective the study drug is at lowering allergic eye signs and symptoms compared with placebo. A placebo looks like a treatment but does not contain any real medicine.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects).

ELIGIBILITY:
Key Inclusion Criteria:

1. Documented or participant-reported history of moderate to severe birch pollen allergy for at least 2 years with bothersome ocular symptoms during the birch season
2. Positive SPT to birch allergen extract, as described in the protocol
3. Positive allergen specific immunoglobulin E (sIgE) tests for birch and Bet v 1 (≥0.7 kUa/L) at screening visit 1
4. Must be able to complete birch screening CACs and meet the criteria, as described in the protocol

Key Exclusion Criteria:

1. Participation in a prior clinical study and received either REGN5713-5714-5715, REGN5713-5715, or REGN5715 antibodies, as described in the protocol
2. Inability to complete or termination of the screening or confirmatory CACs due to a safety concern (eg, anaphylaxis) per Principal Investigator (PI) judgement
3. Significant and/or severe allergies causing symptoms that are expected to coincide or potentially interfere with the study CAC assessments, as assessed by the investigator, as described in the protocol
4. Persistent chronic or recurring acute infection requiring treatment with systemic antibiotics, antivirals, or antifungals, or any untreated respiratory infections within 4 weeks prior to screening visit 1, as described in the protocol
5. The presence of an active ocular infection (bacterial, viral, or fungal) or diagnosis by a physician within 30 days prior to screening visit 1, as described in the protocol

Note: Other protocol defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-08-02 (Actual)

PRIMARY OUTCOMES:
Ocular itch score in response to birch allergen challenge | At Day 8 post-Conjunctival Allergen Challenge (CAC)
  Assessed using the Ora Calibra® Conjunctival Allergen Challenge Ocular Itching Scale, a 0-4 point scale where 0 = none and 4= incapacitating itch, 0.5 unit increments

SECONDARY OUTCOMES:
Conjunctival redness score in response to birch allergen challenge | At Day 8 post-CAC
  Assessed using the Ora Calibra® Hyperemia Scale (for conjunctival [conjunctival redness scale] ciliary [ciliary redness scale], episcleral [episcleral redness scale] vessel beds), a 0 to 4 point scale, where 0 = none and 4 = extremely severe, 0.5 unit increments
Percent change in birch titrated Skin Prick Test (tSPT) in response to birch allergen challenge | Baseline and at Day 8
Tearing score in response to birch allergen challenge | At Day 8 post-CAC
  Assessed using the Ora Calibra® Conjunctival Allergen Challenge Tearing Scale, a 0-4 scale where 0 = none and 4 = very severe, 1 unit increments
Total ocular symptom score (TOSS) in response to birch allergen challenge | At Day 8 post-CAC
  TOSS is a summed score of ocular itch score (graded 0 = none to 4 = incapacitating itch), conjunctival redness score (graded 0 = none to 4 = extremely severe), and tearing score (graded 0 = none to 4 = very severe) for a total range from 0 to 12, where higher scores indicate worse responses.
Total redness score in response to birch allergen challenge | At Day 8 post-CAC
  The total redness score is calculated for CAC: range 0 to 12, where higher scores indicate worse responses (calculated as a sum of the bilateral averages for conjunctival redness score, graded 0 = none to 4 = extremely severe + ciliary redness score, graded 0 = none and 4 = extremely severe + episcleral redness score, graded 0 = none and 4 = extremely severe)
Ciliary redness score in response to birch allergen challenge | At Day 8 post-CAC
  Assessed using the Ora Calibra® Hyperemia Scale (for conjunctival [conjunctival redness scale] ciliary [ciliary redness scale], episcleral [episcleral redness scale] vessel beds), a 0 to 4 point scale, where 0 = none and 4 = extremely severe, 0.5 unit increments
Episcleral redness score | At Day 8 post-CAC
  Assessed using the Ora Calibra® Hyperemia Scale (for conjunctival [conjunctival redness scale] ciliary [ciliary redness scale], episcleral [episcleral redness scale] vessel beds), a 0 to 4 point scale, where 0 = none and 4 = extremely severe, 0.5 unit increments
Change in birch tSPT | Baseline and Day 8
  AUC of the mean wheal diameters
Change in birch tSPT | Baseline and Day 113
  AUC of the mean wheal diameters
Percent change in birch tSPT | Baseline and Day 113
  AUC of the mean wheal diameters
Change in oak tSPT | Baseline and Day 8
  AUC of the mean wheal diameter
Percent change in oak tSPT | Baseline and Day 8
  AUC of the mean wheal diameters
Incidence of Treatment-emergent adverse event (TEAEs) | Up to Day 113
Incidence of serious TEAEs | Up to Day 113
Incidence of Adverse Events of Special Interest (AESIs) | Up to Day 113
Total REGN5713 concentrations in serum over time | Up to Day 113
Total REGN5715 concentrations in serum over time | Up to Day 113
Incidence of Anti-drug antibody (ADAs) to REGN5713 | Up to Day 113
Titers of ADAs to REGN5713 | Up to Day 113
Incidence of ADAs to REGN5715 | Up to Day 113
Titers of ADAs to REGN5715 | Up to Day 113

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (3):
- Andover Eye Associates, Andover, Massachusetts, United States
- Canada (2):
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Clinique de Specialisee en Allergie de la Capitale, Québec

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made results publicly available (e.g., scientific publication, scientific conference, clinical trial registry),
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/